CLINICAL TRIAL: NCT01070134
Title: Mindfulness-based Behavioural Therapy (MIBT) Versus Psychodynamic Therapy for Patients With Major Depressive Disorder in Psychotherapeutic Day Treatment. A Randomised Clinical Pilot Trial
Acronym: Mipsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Psychiatry Roskilde (Industry)
Responsible Party: Janus Jakobsen, Janus Jakobsen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mipsy trial
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-02

CONDITIONS: Major Depressive Disorder; Personality Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Personality Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mindfulness-based Behavioural Therapy (MIBT) (Experimental)
  Interventions: Behavioral: Mindfulness-based Behavioural Therapy (MIBT)
- PT (psychodynamic therapy) (Active Comparator)
  Interventions: Behavioral: PT (psychodynamic therapy)

INTERVENTIONS:
Behavioral: Mindfulness-based Behavioural Therapy (MIBT) — The MIBT treatment consists of weekly individual MIBT therapy (45-50 min.), together with weekly mindfulness-skills training group (1.5 hours).
  The treatment is based on the cognitive model of depression, but will, based on concrete problems, draw from alternative cognitive techniques in order to treat personality-related problems and will use elements from mindfulness.
  Arms: Mindfulness-based Behavioural Therapy (MIBT)
Behavioral: PT (psychodynamic therapy) — The PT treatment consists of weekly individual PT therapy (45-50 min.), together with weekly PT group therapy (1.5 hours).
  The main elements of PT are the free-flowing, non-therapist guided dialogue, based on classic psychoanalytical free association. Basically, the role of the therapist is to set ground rules and organise the time, place and duration, to maintain a proper tone, and ultimately to ensure that a therapeutic process takes place using relevant interventions.
  Arms: PT (psychodynamic therapy)

SUMMARY:
Background:

According to the WHO, major depressive disorder is the second largest healthcare problem worldwide in terms of disability caused by illness. It afflicts an estimated 17% of individuals during their lifetimes at tremendous costs. A number of depressive patients are treated with antidepressant medication. The efficacy of antidepressant medication has been studied in a number of systematic reviews, and in recent years some of these reviews have shown that the efficacy is questionable for many patients. So are there other effective treatments for this serious illness?

Cognitive- and psychodynamic therapies are probably both significantly more effective for depression than no treatment, but only limited comparisons have been made between the two interventions. A Cochrane review shows that cognitive therapy has a preventive effect against recurrent depression, and that this effect may surpass the preventive effect of antidepressant medication. Mindfulness training may be an effective technique in preventing relapse in patients who have had at least 3 previous depressive episodes. But efficacy in treating currently depressed patients has not been studied.

Objective To perform a randomised clinical trial with blinded assessment of efficacy variables in order to study the effects of mindfulness based behavioral therapy (cognitive therapy and mindfulness) versus psychodynamic therapy in depressive patients.

Methods

A randomised clinical trial of 84 consecutive patients diagnosed with major depressive disorder, referred to the day clinic, Roskilde psychiatric services. The patients will be randomised to one of two interventions:

1. MIBT (mindfulness-based behavioural therapy)
2. PT (psychodynamic therapy)

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 65 years
2. Major depressive disorder (SCID I).
3. BDI II > 13.
4. Written informed consent.

Exclusion Criteria:

1. Current psychosis, diagnosis of schizophrenia or schizotypal personality disorder (DSM IV-TR).
2. Alcohol or substance abuse judged to require treatment in preference to depression (assessed during patient conference).
3. Commenced or changed psychopharmacological treatment less than six weeks before randomisation.
4. Pregnancy.
5. No written informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
17 item Hamilton rating scale for depression (score at the end of 18 weeks of day- treatment) | 0 weeks, 18 weeks, and 1 year

SECONDARY OUTCOMES:
SCL-90-R (GSI score at the end of 18 weeks of day- treatment) | 0 weeks, 9 weeks, 18 weeks, and 1 year
The proportion of patients who achieve remission (Hamilton score < 8). | 0 weeks, 18 weeks, and 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- The day clinic for treatment of non-psychotic disorders (Roskilde Psychiatry), Roskilde, Zeeland, Denmark

REFERENCES:
- [Derived] Jakobsen JC, Gluud C, Kongerslev M, Larsen KA, Sorensen P, Winkel P, Lange T, Sogaard U, Simonsen E. Third-wave cognitive therapy versus mentalisation-based treatment for major depressive disorder: a randomised clinical trial. BMJ Open. 2014 Aug 19;4(8):e004903. doi: 10.1136/bmjopen-2014-004903. PMID 25138802
- [Derived] Jakobsen JC, Gluud C, Kongerslev M, Larsen KA, Sorensen P, Winkel P, Lange T, Sogaard U, Simonsen E. 'Third wave' cognitive therapy versus mentalization-based therapy for major depressive disorder. A protocol for a randomised clinical trial. BMC Psychiatry. 2012 Dec 19;12:232. doi: 10.1186/1471-244X-12-232. PMID 23253305